CLINICAL TRIAL: NCT01355744
Title: Swiss Study on Spider Bites
Acronym: SSSB
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SSSB
Record Dates: First submitted 2011-05-17; First posted 2011-05-18 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Spider Bite
Keywords: humans; insect bites
MeSH Terms: conditions — Spider Bites; Insect Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Species of biting spider will be assessed if specimen is sent to us.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spider bite patients: All patients treated for an actual spider bite by a Swiss physician during study period.

SUMMARY:
About spider bites in Middle Europe, there are published only a dozen cases. The investigators suspect that they may be much more frequent than reflected by the literature analysis (but much less dangerous than thought by people). From June 1st 2011 to November 30st 2012 the investigators collect clinical data on patients treated for spider bites in Switzerland.

DETAILED DESCRIPTION:
Inclusion criteria: Every human treated for suspected spider bite in Switzerland willing to participate this study.

ELIGIBILITY:
Inclusion Criteria:

* adult or child treated for a suspected spider bite in Switzerland

Exclusion Criteria:

* unwillingness to participate to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every person with a suspected spider and treated by a Swiss Physician.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Clinical follow up of bite lesions. | 14 days (or more if necessary)
  Clinical evolutions of actual spider bite lesions in humans are observed.

SECONDARY OUTCOMES:
Time spread of spider bites | 18 months
  Frequencies of spider bites over the study period of 18 months are observed.
Causative animals | 18 months
  To determine spider species causing bites in Switzerland by sending spider specimens to an expert arachnologist.

CONTACTS AND LOCATIONS:
Overall Officials: Markus P. Gnädinger, MD, Principal Investigator — Department of General Practice University Hospital Zurich
Locations (1):
- Praxis Dr. med. Markus Gnaedinger, Steinach, Canton of St. Gallen, Switzerland

REFERENCES:
- [Derived] Gnadinger M, Nentwig W, Fuchs J, Ceschi A. Swiss prospective study on spider bites. Swiss Med Wkly. 2013 Sep 4;143:w13877. doi: 10.4414/smw.2013.13877. eCollection 2013. PMID 24019004